CLINICAL TRIAL: NCT05846243
Title: Double-blind, Comparative, Randomized, Placebo-controlled Study on Immunogenicity, Reactogenicity and Safety of Live Cell-based Vaccine Against Smallpox and Other Orthopoxvirus Infections (VACΔ6 Vaccine) in Volunteers Aged 18-60 Years
Brief Title: Study on Immunogenicity, Reactogenicity and Safety of the VACΔ6 Vaccine in Volunteers Aged 18-60 Years
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal Budgetary Research Institution State Research Center of Virology and Biotechnology "Vector" (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VAC∆6-01/20
Record Dates: First submitted 2023-03-23; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-03

CONDITIONS: Smallpox; Monkeypox; Cowpox; Vaccinia Virus Infection
Keywords: VAC∆6 vaccine; Оrthopoxviruses; Smallpox; Сlinical study
MeSH Terms: conditions — Smallpox; Mpox, Monkeypox; Cowpox

STUDY DESIGN:
Intervention Model Description: This was a clinical study of VAC∆6 vaccine designed to induce specific immunity to human-pathogenic orthopoxviruses (VARV, MPXV, CPXV, VACV)
Who Masked: Participant, Investigator
Masking Description: Double-blind Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Group 1 (The first stage): VAC∆6 (10⁷ PFU), Live Smallpox Vaccine (2 months after the vaccination) (Experimental): 15 volunteers aged 18 to 60 who met the inclusion criteria and who received a single intradermal VAC∆6 dose of 1x10⁷ PFU/0.2ml. Live smallpox vaccine was administered by scarification 2 months after the vaccination.
  (The first stage is an open comparative study of the safety, reactogenicity, immunological activity and protective efficacy of VAC∆6 vaccine in two parallel groups).
  Interventions: Biological: VAC∆6 vaccine (10⁷ PFU); Biological: Live Smallpox Vaccine
- Group 2 (The first stage): VAC∆6 (10⁶ PFU), Live Smallpox Vaccine (1 month after the vaccination) (Experimental): 15 volunteers aged 18 to 60 who met the inclusion criteria and who received two intradermal VAC∆6 doses of 10⁶ PFU/0.2ml (given 28 days apart). Live smallpox vaccine was administered by scarification one month after the full vaccination series.
  (The first stage is an open comparative study of the safety, reactogenicity, immunological activity and protective efficacy of VAC∆6 vaccine in two parallel groups).
  Interventions: Biological: VAC∆6 vaccine (10⁶ PFU); Biological: Live Smallpox Vaccine
- Group 3 (The second stage): two intradermal VAC∆6 (10⁶ PFU/0.2 ml) given 28 days apart. (Experimental): 76 volunteers aged 18 to 60 who met the inclusion criteria and who received two intradermal VAC∆6 doses of 10⁶ PFU/0.2 ml (given 28 days apart).
  (The second stage is a Double-blind, Comparative, Randomized, Placebo-controlled study on Immunogenicity, Reactogenicity, and Safety of the VAC∆6 Vaccine in Parallel Groups).
  Interventions: Biological: VAC∆6 vaccine (10⁶ PFU)
- Group 4 (The second stage): two intradermal placebo doses of 0.2 ml (given 28 days apart). (Placebo Comparator): 76 volunteers aged 18 to 60 who met the inclusion criteria and who received two intradermal placebo doses of 0.2 ml (given 28 days apart).
  (The second stage is a Double-blind, Comparative, Randomized, Placebo-controlled study on Immunogenicity, Reactogenicity, and Safety of the VAC∆6 Vaccine in Parallel Groups).
  Interventions: Other: Placebo (Sodium chloride bufus, 0.9%)
- Group 5 (The second stage) in the FGBUZ MSCH-163: a single intradermal VAC∆6 (10⁷ PFU/0.2 ml). (Experimental): 60 volunteers aged 18 to 60 who met the inclusion criteria and who received a single intradermal VAC∆6 dose of 10⁷ PFU/0.2 ml.
  (The second stage is a Double-blind, Comparative, Randomized, Placebo-controlled study on Immunogenicity, Reactogenicity, and Safety of the VAC∆6 Vaccine in Parallel Groups).
  Interventions: Biological: VAC∆6 vaccine (10⁷ PFU)
- Group 6 (The second stage) in the FGBUZ MSCH-163: a single intradermal placebo dose of 0.2 ml. (Placebo Comparator): 60 volunteers aged 18 to 60 who met the inclusion criteria and who received a single intradermal placebo dose of 0.2 ml.
  (The second stage is a Double-blind, Comparative, Randomized, Placebo-controlled study on Immunogenicity, Reactogenicity, and Safety of the VAC∆6 Vaccine in Parallel Groups).
  Interventions: Other: Placebo (Sodium chloride bufus, 0.9%)
- Group 7 (The second stage) in the Hospital No. 1: a single intradermal VAC∆6 (10⁷ PFU/0.2 ml). (Experimental): 16 volunteers aged 18 to 60 who met the inclusion criteria and who received a single intradermal VAC∆6 dose of 10⁷ PFU/0.2 ml.
  (The second stage is a Double-blind, Comparative, Randomized, Placebo-controlled study on Immunogenicity, Reactogenicity, and Safety of the VAC∆6 Vaccine in Parallel Groups).
  Interventions: Biological: VAC∆6 vaccine (10⁷ PFU)
- Group 8 (The second stage): in the Hospital No. 1: a single intradermal placebo dose of 0.2 ml. (Placebo Comparator): 16 volunteers aged 18 to 60 who met the inclusion criteria and who received a single intradermal placebo dose of 0.2 ml.
  (The second stage is a Double-blind, Comparative, Randomized, Placebo-controlled study on Immunogenicity, Reactogenicity, and Safety of the VAC∆6 Vaccine in Parallel Groups).
  Interventions: Other: Placebo (Sodium chloride bufus, 0.9%)

INTERVENTIONS:
Biological: VAC∆6 vaccine (10⁷ PFU) — Live cell-based vaccine against smallpox and other orthopoxvirus infections (VAC∆6 vaccine) based on vaccinia virus (manufactured by FBRI SRC VB "Vector", Rospotrebnadzor).
  Batch: 08-10.19 (expiry date: 13.10.2021). Dosage: single intradermal dose of 10⁷ PFU/0.2 ml of vaccinia virus.
  Arms: Group 1 (The first stage): VAC∆6 (10⁷ PFU), Live Smallpox Vaccine (2 months after the vaccination); Group 5 (The second stage) in the FGBUZ MSCH-163: a single intradermal VAC∆6 (10⁷ PFU/0.2 ml).; Group 7 (The second stage) in the Hospital No. 1: a single intradermal VAC∆6 (10⁷ PFU/0.2 ml).
Biological: VAC∆6 vaccine (10⁶ PFU) — Live cell-based vaccine against smallpox and other orthopoxvirus infections (VAC∆6 vaccine) based on vaccinia virus (manufactured by FBRI SRC VB "Vector", Rospotrebnadzor).
  Batch: 08-10.19 (expiry date: 13.10.2021). Dosage: two intradermal doses of 10⁶ PFU/0.2 ml of vaccinia virus (given 28 days apart).
  Arms: Group 2 (The first stage): VAC∆6 (10⁶ PFU), Live Smallpox Vaccine (1 month after the vaccination); Group 3 (The second stage): two intradermal VAC∆6 (10⁶ PFU/0.2 ml) given 28 days apart.
Biological: Live Smallpox Vaccine — Live smallpox vaccine (Smallpox vaccine) (manufactured by the Federal State Unitary Enterprise NPO Microgen of the Ministry of Health of Russia).
  Batch No. Т30 (expiry date: March, 2021). Dosage: Single 1x10⁶ PFU dose administered by multiple-pricking technique on the 30th/60th day after full series of vaccination with VAC∆6.
  Arms: Group 1 (The first stage): VAC∆6 (10⁷ PFU), Live Smallpox Vaccine (2 months after the vaccination); Group 2 (The first stage): VAC∆6 (10⁶ PFU), Live Smallpox Vaccine (1 month after the vaccination)
Other: Placebo (Sodium chloride bufus, 0.9%) — Sodium chloride bufus, a 0.9% solvent for the preparation of a dosage form for injections (manufactured by JSC Pharmaceutical manufacturing company "Obnovlenie", Russia).
  Batch: 391219 (expiry date: January, 2025).
  Arms: Group 4 (The second stage): two intradermal placebo doses of 0.2 ml (given 28 days apart).; Group 6 (The second stage) in the FGBUZ MSCH-163: a single intradermal placebo dose of 0.2 ml.; Group 8 (The second stage): in the Hospital No. 1: a single intradermal placebo dose of 0.2 ml.

SUMMARY:
The Aim:

Study immunogenicity, confirm the safety and tolerability of different schedules of vaccination with "live cell-based vaccine against smallpox and other orthopoxvirus infections (VAC∆6 vaccine) based on vaccinia virus" using a complex of clinical and laboratory-instrumental techniques.

The research tasks are to:

1. To study the immunological activity of a single VAC∆6 vaccine dose of 1x10⁷ plaque-forming units (PFU).
2. To study the immunological activity of two VAC∆6 vaccine doses (given 28 days apart) of 1x10⁶ PFU.
3. Assess the safety of different VAC∆6 vaccination schedules using a set of clinical and laboratory-instrumental techniques (thermometry, measurement of blood pressure, heart and lung auscultation, ECG, common blood and urine tests, biochemical, immunological and virological studies).
4. Assess the reactogenicity of different VAC∆6 vaccination schedules (number of local and systemic reactions, the percentage of those vaccinated with systemic and local reactions of various severity degrees).
5. To identify VAC∆6 vaccine-associated adverse events.
6. Study cell-mediated immunity induced by different VAC∆6 vaccination schedules.
7. Determine the presence of the virus in specific skin formations (crusts, pustules), saliva, blood and urine.
8. Evaluate the protective efficacy of one and two doses of the studied VAC∆6 vaccine.

DETAILED DESCRIPTION:
This is a Double-blind, Comparative, Randomized, Placebo-controlled Study on Immunogenicity, Reactogenicity and Safety of Live Cell-Based Vaccine Against Smallpox and Other Orthopoxvirus Infections (VAC∆6 Vaccine) Based on Vaccinia Virus in 18-60-year-old Volunteers.

The study included 334 healthy volunteers of both sexes aged 18-60 years who met the inclusion criteria and had no exclusion criteria.

The study was carried out in two stages:

The first stage is an open comparative study of the safety, reactogenicity, immunological activity and protective efficacy of VAC∆6 vaccine in parallel groups of 30 volunteers aged 18 to 60 who met the inclusion criteria. Volunteers were divided into two groups:

* Group 1: 15 volunteers who received a single intradermal VAC∆6 dose of 1x10⁷ PFU. Live smallpox vaccine was administered by scarification 2 months after the vaccination.
* Group 2: 15 volunteers who received two intradermal VAC∆6 doses of 1x10⁶ PFU (given 28 days apart). Live smallpox vaccine was administered by scarification one month after the full vaccination series.

The second stage is a Double-blind, Comparative, Randomized, Placebo-controlled study on Immunogenicity, Reactogenicity, and Safety of the VAC∆6 Vaccine in Parallel Groups. Randomization was carried out using the envelope method. The sealed opaque envelopes included in the Investigator's File were distributed to the clinical sites in the required quantity prior to the start of the study.

Substances were submitted for testing in encrypted form. The encryption technique was chosen and implemented by the sponsor - FBRI SRC VB "Vector", Rospotrebnadzor. Decryption was carried out after study report submission to the Federal Budgetary Research Institution, State Research Center of Virology and Biotechnology "Vector", Rospotrebnadzor.

A total of 304 volunteers aged 18-60 took part in the second stage of the clinical study, of which 158 were men and 146 were women, who met the inclusion criteria and had no exclusion criteria. The volunteers were assigned to study sites as follows:

1. FGBUZ MSCH-163, FMBA Russia - 272 volunteers randomized into four groups:

   * Group 3: 76 volunteers who received two intradermal VAC∆6 doses of 10⁶ PFU/0.2 ml (given 28 days apart);
   * Group 4: 76 volunteers who received two intradermal placebo doses of 0.2 ml (given 28 days apart);
   * Group 5: 60 volunteers who received a single intradermal VAC∆6 dose of 10⁷ PFU/0.2 ml;
   * Group 6: 60 volunteers who received a single intradermal placebo dose of 0.2 ml.
2. State Budgetary Health Institution of the Novosibirsk Region "Municipal Infectious Disease Clinical Hospital No. 1" - 32 volunteers randomized into two groups:

   * Group 7: 16 volunteers who received a single intradermal VAC∆6 dose of 10⁷ PFU/0.2 ml;
   * Group 8: 16 volunteers who received a single intradermal placebo dose of 0.2 ml.

     * Before applying for a state license to the Ministry of the Russian Federation on May 4, 2022, the VACΔ6 vaccine was renamed to OrthopoxVac.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent of a volunteer to participate in a clinical trial obtained prior to any of the study procedures.
2. A verified diagnosis of "healthy" according to standard clinical, laboratory and instrumental methods of examination.
3. Age from 18 to 60 inclusive.
4. Body mass index from 18.5 to 30 kg/m3.
5. Ability to attend all scheduled visits and all scheduled procedures and examinations.
6. Consent of volunteers to use effective methods of contraception throughout the study, including the period of observation for possible post-vaccination reactions.

Exclusion Criteria:

1. Hypersensitivity to any component of the product, allergy to vaccine components.
2. Pregnancy or breastfeeding.
3. The military.
4. Persons in custody in detention facilities and those serving sentences in correctional facilities.
5. Children under 18.
6. Acute infectious or non-infectious diseases, exacerbation of chronic diseases less than 4 weeks prior to the study.
7. Tuberculosis (pulmonary and extrapulmonary).
8. Skin diseases: a) common dermatoses (pemphigus, psoriasis, eczema, atopic dermatitis), including the history of dermatoses; other acute and chronic diseases or impaired skin cover (burns, impetigo, herpes, herpes zoster/chicken pox, pustular diseases).
9. Immunosuppressive conditions: congenital or acquired immunodeficiency syndrome (including HIV infection), leukemia, malignant neoplasms, organ transplantation, cellular and humoral immunodeficiencies.
10. Immunosuppressive therapy: treatment with antimetabolites, high doses of corticosteroids for 14 days or more, radio and x-ray therapy, etc.
11. Regular medication intake less than 2 weeks before the start of the study.
12. Taking immunoglobulin drugs or blood products within the last 3 months before the start of the study.
13. Donation (450 ml of blood or plasma or more) less than 2 months before the start of the study.
14. Cardiovascular diseases: decompensated heart defects, subacute bacterial endocarditis, myocarditis, pericarditis, stage 2-3 hypertension, angina pectoris, myocardial infarction; other forms of pathology: stage 1 hypertension, well-controlled heart defects, angina pectoris (mild forms).
15. Diseases of the kidneys and urinary tract: diffuse glomerulonephritis, congenital nephropathy, chronic renal failure, pyelonephritis, toxic nephropathy (transient).
16. Diseases of the digestive system: cirrhosis of the liver, chronic hepatitis, hepatocerebral dystrophy, acute and chronic pancreatitis, diseases of the biliary tract, gastric ulcer and duodenal ulcer, ulcerative colitis.
17. Diseases of the endocrine system: diabetes mellitus, severe forms of thyrotoxicosis and adrenal insufficiency or dysfunction, thymomegaly, congenital enzymopathy.
18. Systemic connective tissue diseases: systemic lupus erythematosus, discoid lupus, rheumatism, rheumatoid arthritis, systemic vasculitis, systemic scleroderma.
19. Blood diseases: leukemia, Hodgkin's disease, aplastic anemia, hemophilia, Werlhof's disease; hemolytic conditions; deficiency anemia.
20. Allergic diseases: bronchial asthma; asthmatic bronchitis, asthmatic syndrome (associated with a respiratory infection); severe anaphylactic reactions (shock, angioedema of the larynx, etc.) to a variety of food, drug and other allergens; allergic reactions to individual allergens (various rashes, clinical disorders, etc.).
21. Diseases of the ear, throat, nose: chronic tonsillitis and adenoiditis requiring surgical treatment; chronic otitis.
22. Surgery within the previous 2 months.
23. Participation in other clinical trials less than 3 months prior to study enrollment.
24. Persons with alcohol, drug or drug addiction. Drinking more than 10 units of alcohol per week (1 unit of alcohol is equivalent to ½ liter of beer, 200 ml of wine or 50 ml of alcohol) or a history of alcoholism, drug addiction, drug abuse.
25. Mental illness and neurasthenia.
26. Previous treatment with human immunoglobulin preparations, if less than 6 months have passed since the treatment.
27. Failure to meet inclusion criteria.
28. Vaccination with any vaccine less than 2 months prior to study entry.
29. Premenopausal women (last menstrual period ≤ 1 year prior to signing the informed consent) who are not surgically sterile.
30. Women who have reproductive potential and do not use or plan to use approved birth control products throughout the study and do not agree to urine pregnancy testing while participating in the study. Acceptable birth control methods include extrauterine devices, oral, implanted, or injectable contraceptives.
31. Nervous and mental diseases: injuries of the central nervous system (CNS) with residual effects, encephalitis and encephalomyelitis (including post-vaccination), meningitis, polyradiculoneuritis (including the history of polyradiculoneuritis), epilepsy, decompensated or subcompensated hydrocephalus, demyelinating and degenerative lesions of the nervous system (muscle degeneration, etc.), stroke; compensated hydrocephalus, Down's disease, Little's disease, CNS trauma without residual effects, history of febrile convulsions, mental illness.
32. Positive analysis for HIV, viral hepatitis B and C, lues.
33. Other сoncomitant diseases that, in the opinion of the investigator, may interfere with the aims of the study.
34. Serious post-vaccination reactions/complications associated with any previous vaccination.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 334 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Changes in the percentage of vaccinees with a titer of virus-neutralizing antibodies to vaccinia virus ≥1:40, at specified time intervals. | Group 1: at days 1, 30, 60, 89. Groups 2, 3, 4: at days 1, 28, 57, 87, 117. Groups 5, 6, 7, 8: at days 1, 30, 60, 90.
  On control days, the percentage of the vaccinees with a titer of virus-neutralizing antibodies to vaccinia virus ≥1:40 is recorded in the neutralization test in embryonated chicken eggs.
  Value changes of this indicator between time points are assessed.

SECONDARY OUTCOMES:
Change in antibody titers. | Group 1: at days 0, 1, 30, 60, 89. Groups 2, 3, 4: at days 0, 1, 28, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 30, 60, 90.
  Determination of antibody titers to poxviruses using ELISA.
Determination of the lymphocyte migration index (MI) | Group 1: at days 30, 89. Groups 2, 3, 4: at days 1, 28, 57, 117. Groups 5, 6, 7, 8: at days 1, 30, 90.
  Determination of the lymphocyte migration index (MI) is carried out in order to conduct a subsequent assessment of the activity of specific DTH effectors in vitro. The MI is calculated by the formula: MI=A/B, where A is the number of cells in the control wells, B is the number of cells in the experimental wells with an inhibitory dose.
  On control days, the changes in the activity of DTH effectors in vitro is assessed. The assessment of the activity of specific DTH effectors in vitro is carried out according to the MI, which characterizes the migration activity of leukocytes; according to the index of inhibition of migration (MII), which characterizes the intensity of production of lymphokines, and according to the integral indicator of the effector functions (IEF). These MI, MII and IEF for each vaccinated person are compared with the corresponding normal parameters. The reaction is considered positive if the difference between the experimental and control values exceeds 20%.
Determination of the lymphocyte migration inhibition index (MII) | Group 1: at days 30, 89. Groups 2, 3, 4: at days 1, 28, 57, 117. Groups 5, 6, 7, 8: at days 1, 30, 90.
  Determination of the lymphocyte migration inhibition index (MII) is carried out in order to conduct a subsequent assessment of the activity of specific DTH effectors in vitro. The MII is calculated by the formula: MII=B/А, where A is the number of cells in the control wells, B is the number of cells in the experimental wells with an inhibitory dose.
  On control days, the changes in the activity of DTH effectors in vitro is assessed. The assessment of the activity of specific DTH effectors in vitro is carried out according to the migration index (MI), which characterizes the migration activity of leukocytes; according to the MII, which characterizes the intensity of production of lymphokines, and according to the integral indicator of the effector functions (IEF). These MI, MII and IEF for each vaccinated person are compared with the corresponding normal parameters. The reaction is considered positive if the difference between the experimental and control values exceeds 20%.
Determination of the integral indicator of the effector functions (IEF) | Group 1: at days 30, 89. Groups 2, 3, 4: at days 1, 28, 57, 117. Groups 5, 6, 7, 8: at days 1, 30, 90.
  Determination of the integral indicator of the effector functions (IEF) is carried out in order to conduct a subsequent assessment of the activity of specific DTH effectors in vitro. The IEF is calculated by the formula: IEF=С/B, where C is the number of lymphocytes in the test wells with the stimulation dose and B is the number of lymphocytes in the test wells with the inhibitory dose.
  On control days, the changes in the activity of DTH effectors in vitro in each vaccinated person is assessed. The assessment of the activity of specific DTH effectors is carried out according to the migration index (MI), which characterizes the migration activity of leukocytes; according to the index of inhibition of migration (MII), and according to the IEF. These MI, MII and IEF for each vaccinated person are compared with the corresponding normal parameters. The reaction is considered positive if the difference between the experimental and control values exceeds 20%.
Recording the number of local reactions. | Group 1: at days 1-14, 21, 30, 60-74, 80, 89. Group 2: at days 1-14, 21, 28-41, 48, 57, 87-100, 107, 116. Groups 3, 4: at days 1-14, 21, 28-41, 48, 57, 87, 117. Groups 5, 6, 7, 8: at days 1-14, 21, 30.
  On control days, the sum of local reactions is recorded: formation of inoculation elements (redness, swelling and papulo-nodules, pustules, vesicles, erythema, induration). Value changes of this indicator between time points are assessed.
  Evaluation criteria for local reactions:
  1. The intensity or severity of adverse reactions should be assessed on a 4-point scale: 0 - none (no symptoms); 1 - mild (presence of mild symptoms); 2 - medium (symptoms that noticeably impair normal daily activities); 3 - severe (symptoms that interfere with normal daily activities).
  2. The severity of local reactions was assessed according to the following criteria:
     * Hyperemia < 50.0 mm (⌀) or an infiltrate < 25.0 mm (⌀) - weak;
     * Hyperemia ≤ 50.0 mm (⌀) or an infiltrate 26.0-50.0 mm (⌀) - medium;
     * Infiltrate > 50.0 mm (⌀) - strong.
Recording the number of systemic reactions. | Group 1: at days 1-14, 21, 30, 60-74, 80, 89. Group 2: at days 1-14, 21, 28-41, 48, 57, 87-100, 107, 116. Groups 3, 4: at days 1-14, 21, 28-41, 48, 57, 87, 117. Groups 5, 6, 7, 8: at days 1-14, 21, 30.
  Recording the number of systemic reactions (malaise, headache, rise in body temperature, weakness, sweating, sleep and appetite disorders, nausea, vomiting, abdominal pain, etc.). Evaluating criteria for systemic reactions:
  1. The intensity or severity of adverse reactions should be assessed on a 4-point scale: 0 - none (no symptoms); 1 - mild (presence of mild symptoms); 2 - medium (symptoms that noticeably impair normal daily activities); 3 - severe (symptoms that interfere with normal daily activities).
  2. The temperature response should be evaluated according to the following categories in °С: 0 (none) ≤ 37 °C; 1 (weak) > 37 °С - ≤ 37.5 °С; 2 (medium) > 37.5 °С - ≤ 38.5 °С; 3 (strong) > 38.5°C.
Recording of the percentage of the vaccinated with various degrees of manifestation of systemic and local reactions. | Group 1: at days 1-14, 21, 30, 60-74, 80, 89. Group 2: at days 1-14, 21, 28-41, 48, 57, 87-100, 107, 116. Groups 3, 4: at days 1-14, 21, 28-41, 48, 57, 87, 117. Groups 5, 6, 7, 8: at days 1-14, 21, 30.
  Recording of the percentage of the vaccinated with various degrees of manifestation of systemic and local reactions.

OTHER OUTCOMES:
Body temperature monitoring at specified time intervals. | Group 1: at days 0-14, 21, 30, 60-74, 80, 89. Group 2: at days 0-14, 21, 28-41, 48, 57, 87-100, 107, 116. Groups 3, 4: at days 0-14, 21, 28-41, 48, 57, 87, 117. Groups 5, 6, 7, 8: at days 1-14, 21, 30.
  Body temperature is recorded (in degrees Celsius, °C) on control days. The changes in the values of this indicator between time points are assessed.
Arterial blood pressure monitoring at specified time intervals. | Group 1: at days 0-14, 21, 30, 60-74, 80, 89. Group 2: at days 0-14, 21, 28-41, 48, 57, 87-100, 107, 116. Groups 3, 4: at days 0-14, 21, 28-41, 48, 57, 87, 117. Groups 5, 6, 7, 8: at days 1-14, 21, 30.
  Systolic and diastolic blood pressure is recorded (in mmHg). The changes in the values of this indicator between time points are assessed.
Heart rate monitoring at specified time intervals. | Group 1: at days 0-14, 21, 30, 60-74, 80, 89. Group 2: at days 0-14, 21, 28-41, 48, 57, 87-100, 107, 116. Groups 3, 4: at days 0-14, 21, 28-41, 48, 57, 87, 117. Groups 5, 6, 7, 8: at days 1-14, 21, 30.
  The heart rate is recorded (in beats per minute) on control days. The changes in the values of this indicator between time points are assessed.
Monitoring of the frequency of respiratory movements at specified time intervals. | Group 1: at days 0-14, 21, 30, 60-74, 80, 89. Group 2: at days 0-14, 21, 28-41, 48, 57, 87-100, 107, 116. Groups 3, 4: at days 0-14, 21, 28-41, 48, 57, 87, 117. Groups 5, 6, 7, 8: at days 1-14, 21, 30.
  The frequency of respiratory movements (per minute) is recorded on control days. The changes in the values of this indicator between time points are assessed.
Monitoring of the content of erythrocytes (as part of a clinical (general) blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a clinical (general) blood test is performed: the content of erythrocytes (10^12 pcs/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of leukocytes (as part of a clinical (general) blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a clinical (general) blood test is performed: the content of leukocytes (10⁹ pcs/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of hemoglobin (as part of a clinical (general) blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a clinical (general) blood test is performed: the content of hemoglobin (g/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of platelets (as part of a clinical (general) blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a clinical (general) blood test is performed: the content of platelets (10⁹ pcs/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of stab neutrophils (as part of a clinical (general) blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a clinical (general) blood test is performed: the content of stab neutrophils (in %) is measured. The changes in values between time points are assessed.
Monitoring of the content of segmented neutrophils (as part of a clinical (general) blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a clinical (general) blood test is performed: the content of segmented neutrophils (in %) is measured. The changes in values between time points are assessed.
Monitoring of the content of eosinophils (as part of a clinical (general) blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a clinical (general) blood test is performed: the content of eosinophils (in %) is measured. The changes in values between time points are assessed.
Monitoring of the content of basophils (as part of a clinical (general) blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a clinical (general) blood test is performed: the content of basophils (in %) is measured. The changes in values between time points are assessed.
Monitoring of the content of monocytes (as part of a clinical (general) blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a clinical (general) blood test is performed: the content of monocytes (in %) is measured. The changes in values between time points are assessed.
Monitoring of the content of lymphocytes (as part of a clinical (general) blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a clinical (general) blood test is performed: the content of lymphocytes (in %) is measured. The changes in values between time points are assessed.
Erythrocyte sedimentation rate (ESR) monitoring (as part of a clinical (general) blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a clinical (general) blood test is performed: ESR (in mm/h) is measured. The changes in values between time points are assessed.
Monitoring of the enzyme activity of alanine transaminase (as part of a biochemical blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a biochemical blood test is performed: the enzyme activity of alanine transaminase (in U/l) is measured. The changes in values between time points are assessed.
Monitoring of the enzyme activity of aspartate aminotransferase (as part of a biochemical blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a biochemical blood test is performed: the enzyme activity of aspartate aminotransferase (in U/l) is measured. The changes in values between time points are assessed
Monitoring of the enzyme activity of lactate dehydrogenase (as part of a biochemical blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a biochemical blood test is performed: the enzyme activity of lactate dehydrogenase (in U/l) is measured. The changes in values between time points are assessed.
Monitoring of the enzyme activity of alkaline phosphatase (as part of a biochemical blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a biochemical blood test is performed: the enzyme activity of alkaline phosphatase (in U/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of B-lipoproteins (as part of a biochemical blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a biochemical blood test is performed: the content of B-lipoproteins (in mmol/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of cholesterol (as part of a biochemical blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a biochemical blood test is performed: the content of cholesterol (in mmol/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of total protein (as part of a biochemical blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a biochemical blood test is performed: the content of total protein (in g/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of total bilirubin (as part of a biochemical blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a biochemical blood test is performed: the content of total bilirubin (in µmol/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of glucose (as part of a biochemical blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a biochemical blood test is performed: the content of glucose (in mmol/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of creatinine (as part of a biochemical blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a biochemical blood test is performed: the content of creatinine (in µmol/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of urea (as part of a biochemical blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a biochemical blood test is performed: the content of urea (in mmol/l) is measured. The changes in values between time points are assessed.
Monitoring of thymol test (as part of a biochemical blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a biochemical blood test is performed: the thymol test (in S-H units) is measured. The changes in values between time points are assessed.
Monitoring of the content of C reactive protein (CRP) (as part of a biochemical blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a biochemical blood test is performed: the content of CRP (in mg/ml) is measured. The changes in values between time points are assessed.
Monitoring of the prothrombin index (PTI) (as part of a biochemical blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a biochemical blood test is performed: the prothrombin index (in %) is measured. The changes in values between time points are assessed.
Monitoring of the IgE level (as part of a biochemical blood test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a biochemical blood test is performed: the changes in the content of Class E (in IU/ml) immunoglobulins is assessed.
Monitoring of urine transparency (as part of a common urine test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a common urine test is performed: urine transparency is assessed. The changes in urine transparency between time points are assessed.
Monitoring of the specific gravity of urine (as part of a common urine test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a common urine test is performed: the specific gravity of urine is measured. The changes in values between time points are assessed.
Monitoring of the content of protein (as part of a common urine test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a common urine test is performed: the content of protein (in g/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of glucose (as part of a common urine test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a common urine test is performed: the content of glucose (in mmol / l) is measured. The changes in values between time points are assessed.
Monitoring of the content of leukocytes (as part of a common urine test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a common urine test is performed: the content of leukocytes (10⁹/l) is measured. The changes in values between time points are assessed.
Monitoring of the content of erythrocytes (as part of a common urine test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a common urine test is performed: the content of erythrocytes (10^12/l) is measured. The changes in values between time points are assessed.
Monitoring of the casts in urine (as part of a common urine test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a common urine test is performed: the number of casts in the urine is counted (units in the field of view). The changes in values between time points are assessed.
Monitoring of the salts in urine (as part of a common urine test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a common urine test is performed: the number of salt crystals in the urine is counted (crystals per field of view). The changes in values between time points are assessed.
Monitoring of bacteria in urine (as part of a common urine test). | Group 1: at days 0, 1, 5, 14, 30, 60, 66, 73, 89. Group 2: at days 0, 1, 5, 14, 28, 32, 41, 57, 87, 93, 100, 116. Groups 3, 4: at days 0, 1, 5, 14, 28, 31, 41, 57, 87, 117. Groups 5, 6, 7, 8: at days 0, 1, 5, 14, 30, 60, 90.
  On control days, a common urine test is performed: the number of bacteria in the urine is counted (units in the field of view). The changes in values between time points are assessed.
Number of participants with vaccinia virus in blood, urine and saliva. | Groups 3, 4: at days 2-14, 29-41. Groups 5, 6, 7, 8: at days 2-14.
  Оn control days, the determination of the vaccinia virus in blood, urine, and is carried out.
Number of participants with vaccinia virus in specific skin formations (crusts, pustules). | Groups 3, 4: at days 14, 41. Groups 5 - 8: at day 14.
  Оn control days, the determination of the vaccinia virus in specific skin formations (crusts, pustules) is carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir I. Kuzubov, PhD, Principal Investigator — Medical and Sanitary Unit No. 163 (FGBUZ MSCH-163, FMBA Russia) (Novosibirsk); Irina V Krasil'nikova, PhD, Principal Investigator — Municipal Infectious Disease Clinical Hospital No. 1 (Novosibirsk)
Locations (2):
- Russia (2):
  - Federal State Budgetary Institution of Healthcare "Medical and Sanitary Unit No. 163 of the Federal Medical and Biological Agency" (FGBUZ MSCH-163, FMBA of Russia), Kol'tsovo, Novosibirsk Oblast
  - State Budgetary Health Institution of the Novosibirsk Region "Municipal Infectious Disease Clinical Hospital No. 1", Novosibirsk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yakubitskiy SN, Kolosova IV, Maksyutov RA, Shchelkunov SN. Attenuation of Vaccinia Virus. Acta Naturae. 2015 Oct-Dec;7(4):113-21. PMID 26798498
- [Background] Maksyutov RA, Yakubitskyi SN, Kolosova IV, Shchelkunov SN. Comparing New-Generation Candidate Vaccines against Human Orthopoxvirus Infections. Acta Naturae. 2017 Apr-Jun;9(2):88-93. PMID 28740731
- [Background] Olson VA, Shchelkunov SN. Are We Prepared in Case of a Possible Smallpox-Like Disease Emergence? Viruses. 2017 Aug 27;9(9):242. doi: 10.3390/v9090242. PMID 32962316
- [Background] Shchelkunova GA, Shchelkunov SN. Smallpox, Monkeypox and Other Human Orthopoxvirus Infections. Viruses. 2022 Dec 29;15(1):103. doi: 10.3390/v15010103. PMID 36680142
- [Background] Shchelkunova GA, Shchelkunov SN. 40 Years without Smallpox. Acta Naturae. 2017 Oct-Dec;9(4):4-12. PMID 29340212
- [Background] Shchelkunov SN, Shchelkunova GA. Genes that Control Vaccinia Virus Immunogenicity. Acta Naturae. 2020 Jan-Mar;12(1):33-41. doi: 10.32607/actanaturae.10935. PMID 32477596
- [Background] Shchelkunov SN, Shchelkunova GA. [We should be prepared to smallpox re-emergence.]. Vopr Virusol. 2019;64(5):206-214. doi: 10.36233/0507-4088-2019-64-5-206-214. Russian. PMID 32167685
- [Background] Maksyutov RA, Yakubitskiy SN, Kolosova IV, Tregubchak TV, Shvalov AN, Gavrilova EV, Shchelkunov SN. Genome stability of the vaccine strain VACDelta6. Vavilovskii Zhurnal Genet Selektsii. 2022 Jul;26(4):394-401. doi: 10.18699/VJGB-22-48. PMID 35903306
- [Background] Marennikova S.S., Shchelkunov S.N. Orthopoxviruses pathogenic for humans (monograph) // KMK Scientific Press Ltd., M. - 1998, - 386 p (in Russian).
- [Background] Kolosova I.V., Babkina I.N., Yakubitsky S.N., Maksyutov R.A., Safronov P.F., Shchelkunov S.N. Recombinant strain L-IVP 1421ABJCN of vaccinia virus with deleted virulence genes A56R, B8R, J2R, C3L, N1L to obtain a live cell-based attenuated vaccine against smallpox and other orthopoxviruses pathogenic to humans // RF Patent No. 2588388, priority 20.04.2015 (in Russian).
- [Background] Yakubitsky S.N., Kolosova I.V., Maksyutov R.A., Shchelkunov S.N. Recombinant strain VACΔ6 of vaccinia virus with deleted virulence genes C3L, N1L, J2R, A35R, A56R, B8R for obtaining a live cell-based attenuated vaccine against smallpox and other human orthopoxvirus infections // RF Patent No. 2621868, priority 24.06.2016 (in Russian).